CLINICAL TRIAL: NCT02382653
Title: The Analgesic Efficacy of Oral Piroxicam Versus Buccal Fentanyl in Cancer Breakthrough Pain in Patients With Bone Metastases
Brief Title: Oral Piroxicam Versus Buccal Fentanyl in Breakthrough Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Ayman Abd Al-maksoud Yousef, Prof, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 2970/12/14
Record Dates: First submitted 2015-03-03; First posted 2015-03-09 (Estimated); Last update posted 2016-05-13 (Estimated); Status verified 2016-05

CONDITIONS: Neoplasm Metastases
MeSH Terms: conditions — Neoplasm Metastasis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- oral perixicam (Other): 50 patients with Breakthrough pain will receive oral prioxicam for treament of breakthrough pain.
  Interventions: Drug: oral perixicam
- oral fentanyl (No Intervention): 50 patients with Breakthrough pain will receive sublingual fentanyl for treament of breakthrough pain.

INTERVENTIONS:
Drug: oral perixicam — Oral adminstration of buccal perixicam
  Other Names: feldene flash
  Arms: oral perixicam

SUMMARY:
100 patients with Breakthrough pain will be allocated to receive either oral prioxicam (OP) (n=50) or sublingual fentanyl (SLF) (n=50) . Patients will be divided randomly into two equal groups: oral prioxicam (OP) Group and sublingual fentanyl citrate (SLF) Group, comprising of 50 patients each.

Pain intensity level on a 0-10 visual analog scale (VAS), patients will be instructed about the use of a 10-cm visual analog scale (VAS) (0 = no pain to 10 = worst possible pain). frequency of Breakthrough pain throughout the day, onset of relief (0-5, 6-10, 11-15, or over 16 min), time required for dose titration, patient satisfaction and adverse effects were assessed at 3, 7, 15, and 30 days after starting the treatment.

DETAILED DESCRIPTION:
In this prospective, longitudinal, controlled-study, 100 patients with Breakthrough pain will be allocated to receive either oral prioxicam (OP) (n=50) or sublingual fentanyl (SLF) (n=50) . Patients will be divided randomly into two equal groups: oral prioxicam (OP) Group and sublingual fentanyl citrate (SLF) Group, comprising of 30 patients each.

Eligible participants were all adults aged 18 or over suffering from Background pain cancer pain whose cancer pain was treated with strong opioids and who had breakthrough pain which met the criteria described by Portenoy.(5) (stable analgesia in the previous 48 h, controlled background pain in the previous 24 h, transient exacerbation of pain in the previous 24 h). The term strong opioid refers to medicines classified as being on step three of the World Health Organization (WHO) analgesic ladder. In Egypt the strong opioids available include fentanyl, morphine and hydromorphone.

Exclusion criteria were less than18 years old, non-controlled basal pain, hospitalized patients, or cognitive disturbances, patients with contraindication to NSAIDS such as gastric ulcer, impaired renal function, cerebrovascular accident, Coronary artery bypass graft , Uncontrolled hypertension, patients with coagulation anomalies such as hepatic disease or patients a previous history of allergy to NSAID.

Randomization will be performed by random numbers using sealed envelopes without sex stratification. Sealed envelopes indicate the group of assignment. An independent anesthesiologist, who did not participate in the study or data collection, will read the number contained in the envelope and made group assignments. Patients will be blindly randomized to the two groups; the process of inclusion into the study will go on until the requested number of patients will be reached.

Pain intensity level on a 0-10 visual analog scale (VAS), patients will be instructed about the use of a 10-cm visual analog scale (VAS) (0 = no pain to 10 = worst possible pain). frequency of Breakthrough pain throughout the day, onset of relief (0-5, 6-10, 11-15, or over 16 min), time required for dose titration, patient satisfaction and adverse effects were assessed at 3, 7, 15, and 30 days after starting the treatment.

The primary outcome is the degree of breakthrough pain score using VAS in the two groups. The secondary outcomes measures are analgesic requirement, patients satisfaction, and identification of undesirable effects that may be associated with the use of both drugs in patients with breakthrough pain in both groups. All adverse events related to surgery and the regional anesthetic technique will be recorded.

ELIGIBILITY:
Inclusion Criteria:

Eligible participants were all:

* adults aged 18 or over
* suffering from Background pain cancer pain
* whose cancer pain was treated with strong opioids and
* who had breakthrough pain which met the criteria described by Portenoy.

Exclusion Criteria:

Exclusion criteria were:

* less than18 years old,
* non-controlled basal pain,
* hospitalized patients, or cognitive disturbances,
* patients with contraindication to NSAIDS such as:

  * gastric ulcer,
  * impaired renal function,
  * cerebrovascular accident,
  * coronary artery bypass graft,
  * uncontrolled hypertension,
  * patients with coagulation anomalies such as hepatic disease or
  * patients a previous history of allergy to NSAID.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2014-12; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
analgesic scale (assessmet of VAS immeditally after analgesic adminstration) | two hours
  assessmet of VAS immeditally after analgesic adminstration

CONTACTS AND LOCATIONS:
Overall Officials: Ayman A Yousef, Principal Investigator — Assistant professor